CLINICAL TRIAL: NCT06202287
Title: Examining the Relationship Between the Presence of Kinesiophobia in Stroke Patients and Balance, Gait, Pain, and Social Participation Levels
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Furkan Çakır, medical doctor, Ankara City Hospital Bilkent
Other Study IDs: 10026499
Record Dates: First submitted 2024-01-01; First posted 2024-01-11 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Kinesiophobia; Stroke
Keywords: Kinesiophobia; Stroke; balance; pain
MeSH Terms: conditions — Kinesiophobia; Stroke; Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- stroke patient: The specified tests will be administered to 50 patients who have experienced strokes and meet the criteria.
  Interventions: Other: Balance measurements using the HUR Smart balance device, balance tests, and other surveys.

INTERVENTIONS:
Other: Balance measurements using the HUR Smart balance device, balance tests, and other surveys. — 50 stroke patients will undergo balance measurements using the HUR Smart balance device and other tests.

SUMMARY:
The aim of this study is to detect the presence of kinesiophobia, which may affect treatment in stroke patients, and to have an idea about its relationship with kinesiophobia by examining factors such as balance, gait, pain and social participation level.

DETAILED DESCRIPTION:
Individuals aged 18-75 with post-stroke hemiplegia or hemiparesis, a minimum Functional Ambulation Scale score of 2, and no major neurological or rheumatological pathology affecting the musculoskeletal system other than stroke (e.g., Polyneuropathy, Parkinson's, Multiple Sclerosis, Rheumatoid Arthritis, etc.), as well as those without diseases affecting balance (e.g., Parkinson's, Cerebral trauma, Meniere's disease, ear infection, Benign Paroxysmal Positional Vertigo, Multiple Sclerosis), and not using medications that disrupt balance, will be included in the study. Detailed medical histories will be obtained from all included patients and/or caregivers, and comprehensive musculoskeletal examinations will be conducted. Patient information, including name, surname, age, gender, occupation, education level, marital status, body mass index, duration of illness, stroke type, affected side, dominant side, and comorbidities, will be recorded.

All included patients in the study will be assessed by the same physician using the Functional Ambulation Scale, Community Integration Questionnaire , Mini-BESTest (Mini-Balance Evaluation Systems Test), balance assessment on the Hur Smart balance device, The Timed Up and Go Test , Tinetti Balance and Gait Test, Vas Kinesiophobia Scale., and Tampa Kinesiophobia Scale.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18 and 75 years old
* Having experienced post-stroke hemiplegia or hemiparesis
* Scoring at level 2 or above on the Functional Ambulation Classification
* Being willing to participate in the study and signing the consent forms"

Exclusion Criteria:

* Patients who cannot undergo mental evaluation, are unable to complete scales, are illiterate, or have aphasia
* Having major neurological or rheumatological pathologies affecting the musculoskeletal system other than stroke (Polyneuropathy, Parkinson's, Multiple Sclerosis, Rheumatoid Arthritis, etc.)
* Patients with diseases affecting balance (Parkinson's, Cerebral trauma, Meniere's disease, ear infections, Benign Paroxysmal Positional Vertigo, Multiple Sclerosis, etc.)
* Patients using medications that may disrupt balance

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Total of 50 stroke patients meeting the criteria will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2023-10-15 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
The Tampa Scale of Kinesiophobia | baseline
  Scale, "The Tampa Kinesiophobia Scale (TKS) is a self-reported, 17-item scale developed to measure the fear of movement. A high score indicates a high level of fear of movement, while a low score suggests negligible levels of fear of movement.

SECONDARY OUTCOMES:
Visual analogue scale | baseline
  The Visual Analog Scale (VAS) is evaluated on a scale ranging from "no pain" to "worst possible pain." The value of 0 (zero) indicates "no pain," while the value of 10 (ten) indicates "the most severe pain imaginable."
Functional ambulation classification (FAC) | baseline
  Scale, The FAC has six categories ranging from 0 (non-functional ambulation) to 5 (independent). The intermediary categories quantify levels of assistance, supervision, and independent but limited mobility.
Community Integration Questionnaire | baseline
  Questionnaire,The community integration questionnaire (CIQ) was designed to assess home integration, social integration and productive activity in persons with acquired brain injury. The instrument consists of 15 items and can be completed by self report or with the assistance of a family member or caregiver familiar with the person's health status and social activities.
  The community integration questionnaire (CIQ) was designed to assess home integration, social integration and productive activity in persons with acquired brain injury. The instrument consists of 15 items and can be completed by self report or with the assistance of a family member or caregiver familiar with the person's health status and social activities.
Mini-BESTest: Balance Evaluation Systems Test | baseline
  The Mini-BESTest includes four subscales: transitions/anticipatory postural control, reactive postural control, sensory orientation and stability in gait. Each item is rated on a three-point ordinal scale(0 = severe to 2 = normal).The MiniBESTest consists of 14 items, with a maximum score of 28 points
The timed up and go test | baseline
  A 3-meter distance in front of the chair is designated. The patient is asked to stand up from the chair, walk this distance, and then sit down again. The elapsed time provides the result of the test. If the patient takes longer than 12 seconds to complete this test, there is a risk of falling.
Tinetti balance and gait test | baseline
  This test measures the patient's balance and gait ability. The maximum score for the gait component is 12, and for the balance component is 16. The overall maximum score is 28. Generally, patients scoring below 19 are at a high risk of falling.
VAS - Kinesiophobia Assessment | baseline
  To measure motion fear, a Visual Analog Scale was used. A 10-centimeter horizontal line was drawn, ranging from 0 (no fear) at the beginning to 100 (severe fear) at the end. Participants were asked to stand up just before starting exercise and mark the intensity of their motion fear at that moment on the scale.
HUR Smart balance device | baseline
  In the measurement of postural balance parameters, we utilized the HUR SMARTBALANCE BTG4 device and the accompanying software, HUR SmartBalance, available in our clinic. The device, through the balance platform, enables force measurements and load distribution, while sensors detect postural changes. The HUR SmartBalance software within the device provides various balance parameters based on these values, allowing for the assessment of the patient's balance

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital Physical Therapy and Rehabilitation Hospital, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Bak E, Mlynarska A, Marcisz C, Kadlubowska M, Marcisz-Dyla E, Sternal D, Mlynarski R, Krzeminska S. Kinesiophobia in Elderly Polish Patients After Ischemic Stroke, Including Frailty Syndrome. Neuropsychiatr Dis Treat. 2022 Mar 31;18:707-715. doi: 10.2147/NDT.S352151. eCollection 2022. PMID 35387207
- [Background] Wasiuk-Zowada D, Knapik A, Szefler-Derela J, Brzek A, Krzystanek E. Kinesiophobia in Stroke Patients, Multiple Sclerosis and Parkinson's Disesase. Diagnostics (Basel). 2021 Apr 28;11(5):796. doi: 10.3390/diagnostics11050796. PMID 33924856